CLINICAL TRIAL: NCT02999087
Title: A Phase III Randomized Trial of Avelumab-cetuximab-Radiotherapy Versus Standards of Care in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Randomized Trial of Avelumab-cetuximab-radiotherapy Versus SOCs in LA SCCHN (REACH)
Acronym: REACH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2017-01
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HNSCC
Keywords: Head and Neck cancer; Immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Cetuximab; avelumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A Patient FIT (Active Comparator): Lead-in phase (Day-8) : no treatment
  Concomitant radiotherapy phase : Radiotherapy by IMRT + cisplatin 100mg/m2
  Maintenance phase : no treatment until follow-up phase
  Interventions: Drug: Cisplatin; Radiation: IMRT
- Arm B Patient FIT (Experimental): Lead-in phase (Day-8) : Cetuximab 400mg/m2 and avelumab 10mg/kg
  Concomitant radiotherapy phase : Radiotherapy by IMRT + cetuximab 250mg/m2 and avelumab 10mg/kg
  Maintenance phase : avelumab 10mg/kg every 2 weeks during 12 months
  Interventions: Drug: Cetuximab; Drug: avelumab; Radiation: IMRT
- Arm C Patient UNFIT (Experimental): Lead-in phase (Day-8) : Cetuximab 400mg/m2 and avelumab 10mg/kg
  Concomitant radiotherapy phase: Radiotherapy by IMRT + cetuximab 250mg/m2 and avelumab 10mg/kg
  Maintenance phase : avelumab 10mg/kg every 2 weeks during 12 months
  Interventions: Drug: Cetuximab; Drug: avelumab; Radiation: IMRT
- Arm D Patient UNFIT (Active Comparator): Lead-in phase (Day-8): Cetuximab 400mg/m2
  Concomitant radiotherapy phase: Radiotherapy by IMRT + cetuximab 250mg/m2
  Maintenance phase : no treatment until follow-up phase
  Interventions: Drug: Cetuximab; Radiation: IMRT

INTERVENTIONS:
Drug: Cetuximab — Loading dose of 400 mg/m² IV on Day-8, followed by weekly dose of 250 mg/m² IV during the whole course of RT.
  Arms: Arm B Patient FIT; Arm C Patient UNFIT; Arm D Patient UNFIT
Drug: avelumab — IV infusion of avelumab (10 mg/kg over 1 hour) once every 2 weeks. Avelumab will start on Day-8 together with cetuximab and subsequently every 2 weeks during the course of RT. Avelumab with be continued every 2 weeks for an additional 12 months following RT.
  Arms: Arm B Patient FIT; Arm C Patient UNFIT
Drug: Cisplatin — 100 mg/m² IV after hyperhydration and at a maximal rate of 1 mg/min, on days 1, 22, 43.
  Arms: Arm A Patient FIT
Radiation: IMRT — RT will be performed using IMRT (intensity modulated radiotherapy), with a simultaneous integrated boost (SIB) technique. RT dose to the GTV will be 69.96 Gy in 2.12 Gy daily fractions over 6.5 weeks (33 fractions). Prophylactic dose will be 52.8 Gy in 1.6 Gy daily fractions over 6.5 weeks (33 fractions).

SUMMARY:
The purpose of this study is to demonstrate that treatment with avelumab in combination with RT-cetuximab is superior to standard of care (SOC) cisplatin-RT and/or to SOC RT-cetuximab alone in terms of progression-free survival (PFS) in front-line patients with locally advanced SCCHN.

DETAILED DESCRIPTION:
This open-label, randomized, controlled, multicenter phase III study will include 688 patients with LA SCCHN (420 fit for HD cisplatin and 268 unfit for HD cisplatin), histologically confirmed who had not received previous treatment for this setting. The study is designed with the primary objective of demonstrating that treatment with avelumab in combination with cetuximab-RT is superior to SOC Cisplatin-RT or cetuximab-RT alone in terms of PFS. Randomization will assign the 2 treatment arms of each cohort with a 1:1 ratio. In each cohort (fit for cisplatin and unfit for cisplatin), the randomization will be stratified for the 2 most established prognostic factors N stage (N0-N1 vs N2-3) and p16 expression (OPC p16+ versus OPC p16- or non OPC). All patients will be followed until death or at least 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 80 years
2. Performance Status ECOG 0-1
3. Squamous cell carcinoma, previously untreated
4. Stage III, stage IVa (i.e. operable, but not operated) or IVb (non resectable)
5. Oral cavity, oropharynx, hypopharynx or larynx
6. Availability of pre-treatment tumour tissue sample (for p16 & PD -L1 expression, TILs and immune landscape)
7. Recording of alcohol consumption and smoking history
8. Determination of the patient's ability to receive cisplatin 100 mg /m2 for 3 cycles (fit / unfit)*
9. Written informed consent

   * Criteria for determining if a patient is fit for receiving high dose cisplatin:

     * Calculated creatinin clearance ≥ 60 mL/min as determined by the modified. method of Cockcroft and Gault or by the EDTA method
     * Absolute neutrophil count ≥1 500/μL, platelets ≥100 000/μL, hemoglobin ≥ 10 g/dL, aspartate (AST) and alanine transaminase (ALT) less than 2 times the upper limit of the normal range (ULN), total bilirubin ≤ 1.5 mg/dL, serum albumin > 35 g/L
     * Peripheral neuropathy < grade 2
     * No clinical hearing loss (confirmed by audiogram)
     * Cardiac function compatible with hyperhydration; Left ventricular ejection fraction within the institutional normal ranges as measured by echocardiogram

Exclusion Criteria:

1. Nasopharyngeal, paranasal sinuses, nasal cavity tumors or thyroid cancers
2. Squamous cell carcinoma involving cervical neck nodes with unknown primary site
3. Metastatic disease (stage IVc)
4. Viral infection (HIV, Hepatitis B/C)
5. Autoimmune disease
6. Immunodeficiency or immunosuppressive therapy
7. Active CNS disease
8. Interstitial lung disease
9. Active infection
10. Any prior or current treatment for invasive head and neck cancer. This will include but is not limited to: prior tyrosine kinase inhibitors, any monoclonal antibody, induction chemotherapy, prior surgical resection or RT, or use of any investigational agent
11. Weight loss of > 10% during the last 4 weeks (except if renutrition with a feeding tube is planned before the onset of treatment or is ongoing)
12. Concurrent treatment with any other systemic anti-cancer therapy that is not specified in the protocol
13. Concomitant treatment with any drug on the prohibited medication list such as live vaccines
14. History of other malignancy within the last 3 years (exception of in situ carcinoma and skin carcinomas)
15. Significant disease which, in the judgment of the investigator, as a result of the medical interview, physical examinations, or screening investigations would make the patient inappropriate for entry into the trial
16. Known hypersensitivity reaction to study drugs
17. Any social, personal, medical and/or psychological factor(s) that could interfere with the observance of the patient to the protocol and/or the follow-up and/or the signature of the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 74 months
  Time between randomization and the first event among progression (per modified Response Evaluation Criteria in Solid Tumors (RECIST) version v1.1) and death, whatever the cause of death.

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 74 months
Safety: acute adverse events graded by NCI CTCAE v4.03 | From date of randomization to end of study, assessed up to 74 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tao Y, Auperin A, Sun X, Sire C, Martin L, Coutte A, Lafond C, Miroir J, Liem X, Rolland F, Even C, Nguyen F, Saada E, Maillard A, Colin-Batailhou N, Thariat J, Guigay J, Bourhis J. Avelumab-cetuximab-radiotherapy versus standards of care in locally advanced squamous-cell carcinoma of the head and neck: The safety phase of a randomised phase III trial GORTEC 2017-01 (REACH). Eur J Cancer. 2020 Dec;141:21-29. doi: 10.1016/j.ejca.2020.09.008. Epub 2020 Oct 24. PMID 33125944